CLINICAL TRIAL: NCT05248451
Title: The Impact of Chronic Kidney Disease on Risk of Myocardial Injury After Non Cardiac Surgery (MINS). A Retrospective Chart Review.
Brief Title: Chronic Kidney Disease and Myocardial Injury After Non Cardiac Surgery
Acronym: MINS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Su-Yin MacDonell, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H21-00549
Record Dates: First submitted 2022-02-11; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-01

CONDITIONS: Myocardial Injury; Surgery; Chronic Kidney Diseases
Keywords: MINS; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Renal Function: Patients undergoing inpatient non-cardiac surgery at St. Paul's Hospital with normal preoperative Estimated Glomerular Filtration Rate (eGFR) results. eGFR values considered will be from samples drawn within a one year period preceding surgery. Values from samples drawn within the 7 days immediately preceding surgery will be excluded, in order to avoid introducing bias from acute kidney injuries. All available eGFR values in the 7 to 365 days preceding an individual's surgery will be included, and the average of these values will be used as their preoperative eGFR. Investigators will include all people that have one or more measure. Depending on sample size, investigators may decide to limit inclusion to those that have two or more eGFR estimates.
  Interventions: Other: Not an Interventional Study
- Renal Dysfunction, Chronic Kidney Disease (CKD): Patients undergoing non-cardiac surgery with abnormal preoperative Estimated Glomerular Filtration Rate (eGFR). eGFR values considered will be from samples drawn within a one year period preceding surgery. Values from samples drawn within the 7 days immediately preceding surgery will be excluded, in order to avoid introducing bias from acute kidney injuries. All available eGFR values in the 7 to 365 days preceding an individual's surgery will be included, and the average of these values will be used as their preoperative eGFR. Investigators will include all people that have one or more measure. Depending on sample size, investigators may decide to limit inclusion to those that have two or more eGFR estimates. As eGFR is not accurate in the setting of dialysis, patients receiving dialysis for at least 90 days prior to their surgical procedure will also be included as a separate eGFR category.
  Interventions: Other: Not an Interventional Study

INTERVENTIONS:
Other: Not an Interventional Study — Not an Interventional Study

SUMMARY:
Investigators will conduct a retrospective chart review, examining the impact of chronic kidney disease on risk of myocardial injury after non cardiac surgery (MINS). The objective of this study is to examine interactions between preoperative Estimated Glomerular Filtration Rate (eGFR) and the association between preoperative N-Terminal Pro B-Type Natriuretic Peptide (NT-proBNP) and post operative cardiac events in patients undergoing major non cardiac surgery.

DETAILED DESCRIPTION:
In recent years some authors have shown a correlation between increased post operative troponin and increased 30 day mortality in patients with kidney disease that mirrors the known correlation in those with normal renal function. In patients undergoing non cardiac surgery, Walsh et al demonstrated a 4 to 6 fold increased risk of death associated with elevated post operative troponin in patients with reduced (<60 ml/min, but >30ml/min) preoperative estimated glomerular filtration rate (eGFR). A second, more recent study by Liem et al, also found post operative troponin elevations were associated with higher morbidity and mortality risk in patients with chronic kidney disease undergoing non cardiac surgery. Investigators aim to build upon the findings of these authors by examining the relationship between pre operative eGFR, post operative troponin and risk of post operative cardiac events in patients undergoing non cardiac surgery at St Paul's hospital. Investigators will conduct a retrospective chart review of electronic records for all patients undergoing non cardiac, inpatient surgery at St Paul's Hospital from June 1, 2020 to December 31, 2021). Investigators will include all patients for whom preoperative eGFR values are available, and patients on chronic dialysis. Patients are to be stratified by preoperative eGFR and primary outcomes compared between patients with normal vs abnormal preoperative eGFR. Primary outcomes to be reviewed are myocardial injury after non cardiac surgery (MINS) and troponin elevations.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non cardiac surgery, at St Paul's Hospital, during the period spanning June 1 2020 to November 30 2020
* Preoperative eGFR data is available, or chronic dialysis status is known (these patients will not reliably have eGFR measured, and it is not relevant)
* Inpatient surgeries (elective, urgent, and emergent)

Exclusion Criteria:

* Patients undergoing cardiac surgery.
* Patients undergoing day surgery
* Patients for whom Estimated Glomerular Filtration Rate (eGFR) results are not available

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing non cardiac surgery at St Paul's hospital.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-06-22 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial injury after non cardiac surgery (MINS) | Within 30 days post-operatively
  Myocardial injury after non-cardiac surgery (MINS), based on the American Heart Association (AHA) definitions
Troponin Elevation | Postoperative day 1 - 3
  Post-operative high sensitivity Troponin T (hs-TnT) of 20 ng/L to 65 ng/L with an absolute increase of at least 5 ng/L or any concentration > 65 ng/L

SECONDARY OUTCOMES:
Cancellations of elective surgical cases for non-clinical reasons | From June 1, 2020 to December 31, 2021
  Cancellations of elective surgical cases due to COVID-19 implications or staffing issues.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Prabhakar, MD, Principal Investigator — University of British Columbia; Su-Yin MacDonell, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No